CLINICAL TRIAL: NCT05358145
Title: The Training Effects of Tinkering Activities on Cognitive Flexibility in Older Adults From Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); National Taiwan University (Other); National Taiwan Science Education Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 202010050RINB
Record Dates: First submitted 2022-04-06; First posted 2022-05-03 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Training
Keywords: Task-Switching; Electroencephalogram; Cognitive Flexibility; Aging; Brain Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tinkering (Experimental)
  Interventions: Behavioral: Tinkering Activities
- Control Tinkering (Active Comparator)
  Interventions: Behavioral: Control Tinkering Activities
- Board Games (Active Comparator)
  Interventions: Behavioral: Board Games Activities

INTERVENTIONS:
Behavioral: Tinkering Activities — Tinkering activities are activities that comprise elements of science, art, and technology. Through a series of themes objectives, participants can involve interestingly, creatively, and flexibly in the activity when they fulfill the goal with the materials retrievable at the site. Participants will be trained as they involve in the elements hidden within the core of the training, such as problem exploration, active thinking and inference, trial and error, and problem-solving.
  Arms: Tinkering
Behavioral: Control Tinkering Activities — Controlled Tinkering Activities utilize the themes of Tinkering activities but eliminate the core of Tinkering training, hence implementing a new set of activities that emphasize participants strictly follow procedures to complete the similar objective of Tinkering activities. Each participant will end up with a similar piece of work as Tinkering Activities participants would without problem exploration, active thinking and inference, trial and error, and problem-solving.
  Arms: Control Tinkering
Behavioral: Board Games Activities — Board games are often constructed with concepts of different cognitive components, such as attention, working memory, planning, calculation; therefore serve as a commonly seen cognitive training, while more and more literature continues to support tabletop games being the medium of cognitive promotion.
  Arms: Board Games

SUMMARY:
Aging has been a serious global-wise concern in public health. In particular, elders face declination of cognitive functions that threaten their quality of life. A good approach to slow down cognitive declination during aging processes is therefore in urgent need. According to the Successful Aging model (Rowe, J.W. and Kahn, R.L) participation in meaningful occupational activity may maintains high cognitive and body function. This sub-project is a part of the larger integrated project that will address the need for cognitive promotion by conducting cognitive training interventions on community older adults, utilizing the National Taiwan Science Education Center (NTSEC) as the public recruiting site as well as intervention site. In this sub-project, a 12-week intervention will be carried out with three protocols: 1) Tinkering activities, 2)Controlled Tinkering Activities, and 3) Board Game intervention. Board games serve as a commonly seen cognitive training, with a growing series of literature continuing to support board games being the medium of cognitive promotion. Tinkering activities are primarily used in fields of education that comprise science, art, and technology. Through a series of themes objectives, participants can involve interestingly, creatively, and flexibly in the activity when the participants fulfill the goal with the materials retrievable at the site. The anticipation is that the elders participating in Tinkering activities may increase their cognitive flexibility as the participants involve in the elements hidden within the core of the training, such as problem exploration, active thinking and inference, trial and error, and problem-solving. The investigators target to obtain pre-and post-intervention behavioral and neurophysiological data, including electroencephalogram data in 40 experimental participants, 40 active control participants, and 40 passive control participants over a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Literate in Mandarin and Taiwanese
* Willing to participate entirely in this research.
* Age >65

Exclusion Criteria:

* Participated in cognitive-related training in the past two months.
* Severe impairment of visual or auditory abilities.
* Diagnosed with mild cognitive impairment (MCI), or Dementia
* Severe psychological or behavioral disorder that would seriously interfere with the progress of activity
* History of degenerative cognitive disorder (e.g., acute stroke, traumatic brain injury, unconscious), organic mental disorders, brain dysfunction, or other neurology-related diagnoses.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 118 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Changes of Event-related potential component (ERP): P2, N2, P3 | Week 0, Week 12, Week 36
  The EEG data is recorded while the participants are carrying out the task-switching paradigm. The data will then be analyzed in terms of Event-Related Potential(ERP), where the components' changes will be observed in terms of amplitude and latency.
Changes of reaction time and accuracy of task-switching paradigm | Week 0, Week 12, Week 36
  The task-switching paradigm will ask the participants to judge whether the number(stimulus) presented is 1) even or odd, OR, 2) more than or less than 5. The switching between these rules will induce a switch cost effect (the time when the rule changes, the reaction time will increase to compensate the cognitive process needed to make the change) if the reaction time decreases after intervention, it implies an improvement.
Changes of Accuracy in Wisconsin Card Sorting Test | Week 0, Week 12, Week 36
  Score ranged 0-128, the higher the score, the better the executive function
Changes of Number of Categories Completed in Wisconsin Card Sorting Test | Week 0, Week 12, Week 36
  The number of sequences of 10 consecutive correct matches (maximum = 6), higher the score, the better the executive function
Changes of Trials to Complete First Category in Wisconsin Card Sorting Test | Week 0, Week 12, Week 36
  Total number of trials to complete first category, the less the score, the better the executive function
Changes of Percent Perseverative Errors in Wisconsin Card Sorting Test | Week 0, Week 12, Week 36
  The concentration of perseverative errors in relation to overall test performance (the number of trials given) multiplied by 100. The less the score, the better the executive function.
Changes of Failure to Maintain Set in Wisconsin Card Sorting Test | Week 0, Week 12, Week 36
  When a participant makes five or more consecutive correct matches but then makes an error before successfully completing the category, the less the score, the better the executive function.

SECONDARY OUTCOMES:
Changes of University of California, Los Angeles Loneliness Scale | Week 0, Week 12, Week 36
  score ranged 20-80, the higher the greater sense of loneliness in the participants.
Changes of Geriatric Depression Scale | Week 0, Week 12, Week 36
  Score ranged 0-15, the higher the score, the severe the depressive symptoms.
Changes of Flow Scale | Week 0, Week 12, Week 36
  Score ranged 1-5, higher the score, the better the flow experience the participant had.
Changes of Cognitive Flexibility Scale (CFS) | Week 0, Week 12, Week 36
  It is a 12-item 6-point scale in Likert format, the higher the score, the higher the participants' cognitive flexibility.
Changes of Guilford's Alternative Uses Test (GAU) | Week 0, Week 12, Week 36
  Scoring in terms of originality, fluency, elaboration and flexibility. The higher the score the better the creativity and divergent thinking.
Changes of Color Trails Test (CTT) | Week 0, Week 12, Week 36
  Measures in time, error, cues, near miss, and color error. The less time, error, cues, near miss and color error the participants take, the better the executive function, alternate and sustain attention.
Changes of University of California, San Diego Performance-Based Skills Assessment (UPSA-BRIEF) | Week 0, Week 12, Week 36
  Score range 0-100, the higher the score, the better the function of activities of daily living.
Changes of Remote Associates Test | Week 0, Week 12, Week 36
  Score range 0-30. The higher the score, the better the ability of remote associate creativity.
Changes of Neural functional activity during inferential processing | Week 0, Week 12
  Participants will undergo a Rule Inference functional magnetic resonance imaging task to infer underlying rules that map color configurations of circles in a triangular arrangement to a target color category within as few tries as possible under active or passive conditions. The goal for participants will be to infer the cue-category association rules using as few cues as possible. The primary outcome measure here is the degree of neural response estimate change in blood oxygen level dependent (BOLD) signal pre- and post-intervention.
Changes of overall accuracy during inferential processing | Week 0, Week 12
  Changes from pre- to post-intervention in participant overall accuracy in identifying latent rules in the Rule Inference functional magnetic resonance imaging task.
Changes of learning rate during inferential processing | Week 0, Week 12
  Changes from pre- to post-intervention in participant number of trials to criterion in the Rule Inference functional magnetic resonance imaging task.
Changes of strategic performance during inferential processing | Week 0, Week 12
  Changes from pre- to post-intervention in participant coefficients of expression of modeled response strategies in the Rule Inference functional magnetic resonance imaging task will be assessed.
Change in Wechsler Memory Scale III Logical Memory I & II | Week 0, Week 12
  Score range 0 - 75. Higher score indicates better verbal episodic memory.
Change in Wechsler Memory Scale III Face Memory | Week 0, Week 12
  Score range 0 - 48. Higher score indicates better visual face memory.
Change in Wechsler Memory Scale III Verbal Paired Memory | Week 0, Week 12
  Score range 0 - 32. Higher score indicates better verbal memory and learning.
Change in Wechsler Memory Scale III Family Pictures I & II | Week 0, Week 12
  Score range 0 - 64. Higher score indicates better visual memory and learning.
Change in Wechsler Memory Scale III Word Lists I & II | Week 0, Week 12
  Score range 0 - 36. Higher score indicates better verbal memory and learning. For II, recall score range is 0 to 8; recognition score range is 0 to 24.
Change in Wechsler Memory Scale III Visual Reproduction I & II | Week 0, Week 12
  Score range 0 - 104. Higher score indicates better visual memory. For II, recall score range is 0-104; recognition score range is 0-48.
Change in Wechsler Memory Scale III Spatial Span | Week 0, Week 12
  Score range 0 - 32. Higher score indicates better spatial memory.
Change in Wechsler Memory Scale III Digit Span | Week 0, Week 12
  Score range 0 - 32. Higher score indicates better auditory memory.
Change in Wechsler Adult Intelligence Scale III Vocabulary | Week 0, Week 12
  Score range 0 - 66. Higher score indicates better vocabulary.
Change in Wechsler Adult Intelligence Scale III Digit Symbol | Week 0, Week 12
  Score range 0 - 133. Higher score indicates better processing speed.
Change in Wechsler Adult Intelligence Scale III Block Design | Week 0, Week 12
  Score range 0 - 68. Higher score indicates better visual processing.
Change in Wechsler Adult Intelligence Scale III Arithmetic | Week 0, Week 12
  Score range 0 - 22. Higher score indicates better mathematical computation ability.
Change in Wechsler Adult Intelligence Scale III Matrix Reasoning | Week 0, Week 12
  Score range 0 - 26. Higher score indicates better reasoning.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Fen Mao, M.S., Principal Investigator — National Taiwan University
Locations (2):
- Taiwan (2):
  - College of Medicine, National Taiwan University, Taipei
  - National Taiwan Science Education Center, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Data that can be shared include anonymized neuropsychological assessment scores, cognitive behavioral performance scores, brain imaging data that have been published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available 1 year after primary results are published by the central research team. Data are anticipated to be available for sharing for an indefinite period after the above criteria is met.
Access Criteria: Data sharing will be done based direct requests and on case-by-case evaluation for appropriateness. Use of shared data will require agreement on appropriate citation of data sources at least or authorship inclusion or acknowledgement.